CLINICAL TRIAL: NCT05009030
Title: Observational Study on the Effectiveness and Safety of Vaccination Anti-SARS-CoV2 in Patients With Lung Cancer
Brief Title: Anti-SARS-COV2 Vaccination Study in Lung Cancer Patients
Acronym: VAC-CaP
Status: Completed | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 21/01_VAC-CaP
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Lung Cancer; Covid19
Keywords: COVID-19 vaccine
MeSH Terms: conditions — Lung Neoplasms; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with lung cancer of any histology and stage who receive an anti-COVID-19 vaccine approved by the health authorities. Patients would be eligible whether they have suffered from SARS-CoV2 infection or have not had COVID19.
  Interventions: Drug: COVID-19 vaccine

INTERVENTIONS:
Drug: COVID-19 vaccine — Lung cancer patients will receive an anti-COVID19 vaccine approved by the European Medicines Agency according to the guidelines approved by the regulatory authorities

SUMMARY:
Observational and multicenter retrospective study of data collection in hospital centers throughout the Spanish geography.

This study aims to be nationwide in order to study general common variables of the patients, as well as the correlation with the cancer treatments received.

DETAILED DESCRIPTION:
Observational and multicenter retrospective study of data collection in hospital centers throughout the Spanish geography.

This study aims to be nationwide in order to study general common variables of the patients, as well as the correlation with the cancer treatments received.

Disease and study population Patients with lung cancer of any histology and stage who receive an anti-COVID-19 vaccine approved by the health authorities. Patients would be eligible whether they have suffered from SARS-CoV2 infection or have not had COVID19.

The study will be extended to all the centers of the Spanish Lung Cancer Group, more than 170 centers and 500 professionals, and it is expected that around 500 cases will be collected.

The main objective of the study is to collect the safety and efficacy of the vaccine against SARS-CoV-2 in cancer patients, as well as its potential interactions with antineoplastic therapies.

The data collection will take place throughout the year 2021

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with lung cancer of any stage and histology who have or have not contracted COVID-19 and who have been vaccinated with an EMA approved COVID-19 vaccine.
* Age equal to or greater than 18 years

Exclusion Criteria:

* Patients who have not received an EMA approved COVID-19 vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer of any histology and stage who receive an anti-COVID-19 vaccine approved by the health authorities. Patients would be eligible whether they have suffered from SARS-CoV2 infection or have not had COVID19.
Sampling Method: Non-Probability Sample
Enrollment: 794 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of the COVID19 vaccine | From the date of the last dose of the vaccine until three months later
  Analyze patients who do not become infected with COVID-19 after being vaccinated
Incidence of COVID-19 vaccine-Emergent Adverse Events (Safety and Tolerability) | From the date of first dose of COVID-19 vaccine through 90 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Determine the frequency of COVID-19 and its severity in lung cancer patients receiving the anti-COVID vaccine | From the date of the last dose of the vaccine until three months later
  Analyze patients who become infected with COVID-19 after being vaccinated
Incidence of COVID-19 vaccine-Emergent Adverse Events and toxicities associated with antineoplastic treatments (Safety and Tolerability) | From the date of first dose of COVID-19 vaccine through 90 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Nadal, MD, Study Chair — Fundación GECP Investigator
Locations (51):
- Spain (51):
  - Complejo Hospitalario Universitario De Santiago, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital De Torrevieja, Torrevieja, Alicante
  - Hospital Universitario Araba-Sede Txagorritxu, Vitoria-Gasteiz, Araba
  - Hospital Germans Trias I Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital De Mataro, Mataró, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao, Bizkaia
  - Hospital La Mancha Centro, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Jerez De La Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital San Pedro De Logroño, Logroño, La Rioja
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario De Mostoles, Móstoles, Madrid
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Verge De La Cinta, Tortosa, Tarragona
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Hospital Universitario De A Coruna, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Nuestra Señora De Sonsoles, Ávila
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de Basurto, Bilbao
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Hospital San Cecilio, Granada
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Fundación de Alcorcón, Madrid
  - Hospital General Universitario de Málaga, Málaga
  - Hospital Universitari Son Llatzer, Palma de Mallorca
  - Complejo Hospitalario Pontevedra, Pontevedra
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora La Candelaria, Santa Cruz de Tenerife
  - Hospital General De Segovia, Segovia
  - Hospital De Valme, Seville
  - Hospital De Sant Pau i Sta. Tecla, Tarragona
  - Hospital Virgen De La Salud, Toledo
  - Instituto Valenciano De Oncología, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid
  - Complejo Asistencial De Zamora, Zamora
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org